CLINICAL TRIAL: NCT04622085
Title: The Evaluation of the Safety and Effectiveness of ANIMERS Chiara LA and JUVÉDERM VOLUMA® for Aging Mid-Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDCT-AHSK
Record Dates: First submitted 2020-10-18; First posted 2020-11-09 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Dermal Filler; Hyaluronic Acid; Lidocaine; Aging Mid-Face

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANIMERS Chiara LA (Experimental)
  Interventions: Device: ANIMERS Chiara LA
- JUVÉDERM VOLUMA® (Active Comparator)
  Interventions: Device: JUVÉDERM VOLUMA®

INTERVENTIONS:
Device: ANIMERS Chiara LA — 20mg/SciVision Biotech Inc.
  Arms: ANIMERS Chiara LA
Device: JUVÉDERM VOLUMA® — 20mg/Allergan, Inc.
  Arms: JUVÉDERM VOLUMA®

SUMMARY:
This study is to evaluate the safety and effectiveness for the correction of aging mid-face of treatment group compared with the active control group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 to 60 years of male or female
2. MidFace Volume Deficit Scale (MFVDS) of midface graded 2 to 5 by evaluator.

Exclusion Criteria:

1. Injection site with infection or other skin diseases present which may affect the evaluation
2. With medical history of chromatosis, discoloration, keloid formation, hypertrophic scarring at midface
3. With permanent implants or planning to receive permanent implants during the study period at the injection sites
4. Hyaluronate facial dermal implant injection or other impermanent dermal fillers injection at injection sites within the past 6 months
5. With under-eye facial Botox or fat injection within the past 6 months or planning to receive under-eye facial Botox or fat injection during the study period
6. With Major surgery 3 months before the start of the trial
7. With under-eye facial chemical or lasers peeling, non-invasive skin tightening, thermocool within the past 3 months or planning to receive these aesthetic procedures during the study period
8. With systemic immunosuppressive therapy or systemic corticosteroids within the past 2 months or planning to receive these therapies during the study period (subjects who have received inhaled/intranasal corticosteroids could be considered to include.)
9. With clinical meaningful coagulation disorders, underdoing anticoagulant treatment or within the past 10 days, or taking blood circulation promotion and blood stasis movement medications
10. With epilepsy or porphyria
11. With congenital or idiopathic methemoglobinemia or glucose-6-phosphate dehydrogenase deficiency
12. With analgesic dependence, analgesics within the past 2 weeks or planning to receive analgesics during the study period
13. With history of hypersensitivity or allergy to lidocaine, amide anesthetics, hyaluronic acid or any component of the device; Gram-positive bacterial or Streptococcus proteins; other severe hypersensitivity history unsuitable for participating in the study
14. Planning to undergo any surgery which may cause significant body weight change (such as bariatric surgery) or take any medication which may cause significant body weight change
15. Pregnant, planning pregnancy or in breastfeeding females
16. Participated in clinical study of other device or drug and have not terminated within the past 30 days -Other circumstances which judged to be unsuitable for participating in the study by the investigator

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Response rate of a ≥ 1 Grade improvement on the assessment of MidFace Volume Deficit Scale (MFVDS) | 6 months post-injection
  The response rate is ≥ 1 Grade improvement on the assessment of MidFace Volume Deficit Scale (MFVDS) as assessed by the evaluator at 6 months.
  Evaluators assess the midface volume deficit scale (MFVDS) on site with 5 graded scale, 0 to 5 was represented 'Fullness' to 'Severe concavity'.

SECONDARY OUTCOMES:
Face fullness value evaluated by the digital image scoring system after injection and post 1, 3, 6, 12, 18, 24 months. | Immediate, 1, 3, 6, 12, 18 and 24 months post-injection
  The digital image scoring system analyzes the volume change (ml). A higher score means more volume increased in the midface.
MFVDS value evaluated by blinded-evaluator after injection and 1, 3, 6, 12, 18, 24 months. | Immediate, 1, 3, 6, 12, 18 and 24 months post-injection
  Evaluators assess the midface volume deficit scale on site with 5 graded scale, 0 to 5 was represented 'Fullness' to 'Severe concavity'.
A Response rate of MFVDS value evaluated by blinded-evaluator after injection and 1, 3, 6, 12, 18, 24 months. | Immediate, 1, 3, 6, 12, 18 and 24 months post-injection
  The response rate is ≥ 1 Grade improvement on the assessment of the MidFace Volume Deficit Scale (MFVDS) as assessed by the evaluator after injection and 1, 3, 6, 12, 18, 24 months.
  Evaluators assess the midface volume deficit scale (MFVDS) on site with 5 graded scale, 0 to 5 was represented 'Fullness' to 'Severe concavity'.
GAIS evaluated photographically by blinded-evaluator after injection and 1, 3, 6, 12, 18, 24 months. | Immediate, 1, 3, 6, 12, 18 and 24 months post-injection
  Evaluators and subjects assess the improvement of correction with 5 graded scale,1 to 5 was represented 'exceptional improvement' to 'worsened'.
VAS pain evaluated immediately and 15, 30, 45 and 60 minutes after injection | Immediate,15, 30, 45 and 60 minutes post-injection
  The VAS scale uses a 100 mm line labelled at '0' with 'no pain' and '100' with 'worst pain'.
Adverse events reported during the study period | Immediate, 1, 3, 6, 12, 18 and 24 months post-injection
  The safety assessment was based on reports of adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded during each follow up and at any time the patient reported an event to the investigator during the study period.
Serious adverse events reported during the study period | Immediate, 1, 3, 6, 12, 18 and 24 months post-injection
  The safety assessment was based on reports of adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded during each follow up and at any time the patient reported an event to the investigator during the study period.
Device failure reported before injection | Before injection
  The safety assessment was based on reports of adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded during each follow up and at any time the patient reported an event to the investigator during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan